CLINICAL TRIAL: NCT05405309
Title: A Phase Ib/II Trial of Combination RP-3500 and Olaparib in DNA Damage Repair Pathway Deficient Relapsed/Refractory Chronic Lymphocytic Leukemia
Brief Title: RP-3500 and Olaparib in DNA Damage Repair Pathway Deficient Relapsed/Refractory Chronic Lymphocytic Leukemia
Acronym: CORONADO CLL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to sponsor de-activation of all programs associated with RP-3500 (camonsertib).
Sponsor: University of Utah (Other)
Collaborators: Repare Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCI141431
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase Ib: Dose Level -1 (Experimental): To assess the MTD of RP-3500 in combination with olaparib. Patients will receive RP-3500 40mg daily and olaparib 100mg BID. Both drugs are given with intermittent dosing of 2 days per week and each cycle is 21 days.
  Interventions: Drug: RP-3500; Drug: Olaparib
- Phase Ib: Dose Level 1 (Experimental): To assess the MTD of RP-3500 in combination with olaparib. Patients will receive RP-3500 50mg daily and olaparib 100mg BID. Both drugs are given with intermittent dosing of 2 days per week and each cycle is 21 days.
  Interventions: Drug: RP-3500; Drug: Olaparib
- Phase Ib: Dose Level 2 (Experimental): To assess the MTD of RP-3500 in combination with olaparib. Patients will receive RP-3500 80mg daily and olaparib 100mg BID. Both drugs are given with intermittent dosing of 2 days per week and each cycle is 21 days.
  Interventions: Drug: RP-3500; Drug: Olaparib
- Phase Ib: Dose Level 3 (Experimental): To assess the MTD of RP-3500 in combination with olaparib. Patients will receive RP-3500 80mg daily and olaparib 150mg BID. Both drugs are given with intermittent dosing of 2 days per week and each cycle is 21 days.
  Interventions: Drug: RP-3500; Drug: Olaparib
- Phase II: Dose Expansion Enrichment Cohort (Experimental): Subjects enrolled into the enrichment cohort must have a del(11q) and/or ATM mutation.
  Interventions: Drug: RP-3500; Drug: Olaparib
- Phase II: Dose Expansion Eligible Subjects Cohort (Experimental): Cohort will include all other eligible subjects for Dose Expansion.
  Interventions: Drug: RP-3500
- Phase Ib (prior to Aug2023 amendment): Original Dose Level 1 (Experimental): To assess the MTD of RP-3500 in combination with olaparib. Before the Aug2023 amendment, patients enrolled at Dose Level 1 received RP-3500 40mg daily and olaparib 100mg BID. Both drugs were given with intermittent dosing of 3 days per week and each cycle was 28 days.
  Interventions: Drug: RP-3500; Drug: Olaparib

INTERVENTIONS:
Drug: RP-3500 — RP-3500 is a highly potent and selective Ataxia telangiectasia and Rad3 related inhibitor (ATRi) and has demonstrated significant preclinical activity.
Drug: Olaparib — Olaparib is an oral poly (adenosine diphosphate-ribose) polymerase inhibitor (PARPi) that inhibits PARP's function by competitively binding to the Nicotinamide adenine dinucleotide (NAD+) binding site, which PARP requires as a cofactor to operate.
  Arms: Phase II: Dose Expansion Enrichment Cohort; Phase Ib (prior to Aug2023 amendment): Original Dose Level 1; Phase Ib: Dose Level -1; Phase Ib: Dose Level 1; Phase Ib: Dose Level 2; Phase Ib: Dose Level 3

SUMMARY:
This is an open-label, multicenter, phase Ib/II study of the combination of RP-3500 and olaparib in Relapsed/Refractory Chronic Lymphocytic Leukemia (R/R CLL) patients with DDR deficiencies.

DETAILED DESCRIPTION:
The Phase Ib part of the trial will seek to assess the Maximum Tolerated Dose (MTD) of camonsertib (RP-3500) in combination with olaparib. Given the potential overlapping toxicities of RP-3500 and olaparib, a keyboard phase I design, a novel Bayesian method that typically underestimates the MTD,61 will be employed. The target toxicity is 30% with an equivalence interval between 25-33% of patients. With an anticipated 3 dose levels (DL) and an option for a DL-1, up to 18 patients may be required to determine the MTD. A maximum of 12 patients will be treated at a DL.

The first 5 patients treated at the previous DL1 (camonsertib 40mg daily and olaparib 100mg two times a day (BID) dosing 3 days per week) determined that this dosing strategy may not be appropriate for R/R CLL patients and reduced dosing may be necessary to increase safety of the combination therapy. Therefore, the newly proposed DLs will seek to enroll an additional 18 patients.

After completion of the phase Ib portion and assignment of the recommended phase 2 dose (RP2D), continuous enrollment of patients may commence into the phase II dose expansion portion. All patients enrolled at the RP2D during the phase Ib dose-escalation portion of the trial can be carried over into the phase II analysis. The maximum number of patients that can be carried over from the dose escalation to the dose-expansion portion is 12.

The phase II dose expansion will consist of two separate cohorts of subjects: an enrichment cohort and a cohort for all other eligible subjects. All subjects enrolled into the enrichment cohort must have a del(11q) and/or ATM mutation. Eight subjects will be enrolled into the enrichment cohort and 16 will be enrolled into the second cohort for a total phase II cohort of 24 patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic lymphocytic leukemia (CLL) according to the National Cancer Institute International Workshop on Chronic Lymphocytic Leukemia (NCI/IWCLL), criteria.

  --This includes previous documentation of:
  * Biopsy-proven small lymphocytic lymphoma/CLL
  * OR
  * Diagnosis of CLL according to the NCI/IWCLL criteria as evidenced by all of the following:

    * Peripheral blood monoclonal B cell population of greater than 5x109/L
    * Immunophenotype consistent with CLL defined as:

      * The predominant population of lymphocytes share both B cell antigens [CD19, CD20 (typically dim expression), or CD23] as well as CD5 in the absence of other pan-T-cell markers (CD3, CD2, etc).
      * Clonality as evidenced by κ or λ light chain restriction (typically dim immunoglobulin expression)
  * Negative Fluorescence in situ hybridization (FISH) analysis for t(11;14)(IgH/CCND1) on peripheral blood or tissue biopsy (e.g. marrow aspirate), or negative immunohistochemical stains for cyclin D1 on involved tissue biopsy (e.g. marrow aspirate or lymph node biopsy).
* Repeat testing of somatic mutations and FISH analysis must be performed by a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory after progression is noted from most recent line of therapy and within 6 months of screening. Primary CLL cells must harbor one of these abnormalities:

  * Somatic gene mutation testing shows mutation(s) in Tumor protein P53 (TP53), Ataxia-telangiectasia mutated (ATM), Splicing factor 3b subunit 1 (SF3B1), eukaryotic nuclear export protein exportin-1 (XPO1) and/or Protection of Telomeres Protein 1 (POT1)
  * Cytogenetic FISH analysis shows deletion 17p13 and/or deletion 11q22.3
* Relapsed or refractory after at least 2 prior lines of therapy, and in the opinion of the treating Investigator are either not eligible for other approved therapies or no approved therapies are expected to have sustained therapeutic benefit.
* Patient in need of treatment or change in treatment per iwCLL criteria.

  --Patients on Bruton tyrosine kinase (BTK), Phosphoinositide 3-kinase inhibitor (PI3K) or B-cell lymphoma 2 (BCL2) inhibitors may enroll without meeting iwCLL criteria for treatment as long as there is clinical evidence of progression (i.e. increasing lymphocytosis, worsening anemia/thrombocytopenia attributable to CLL disease progression, increasing lymphadenopathy, or worsening patient symptoms) and require change in treatment at the discretion of the treating provider. Patients must still meet all other inclusion/exclusion criteria for enrollment including appropriate washout periods (5.2.2) and relapsed disease after 2 prior lines of therapy with no other approved therapies that are expected to have sustained therapeutic benefit (5.1.3).
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status between 0-2
* Expected life expectancy of at least 12 months per the investigator.
* The following laboratory or clinical values obtained ≤ 42 days prior to enrollment:

  * Absolute neutrophil count ≥1000/µL (G-CSF support is allowed) unless documented bone marrow involvement of CLL
  * Platelets of ≥50K/µL unless documented bone marrow involvement of CLL
  * Creatinine Clearance (CrCl) ≥45 mL/minute as measured by a 24 hour urine collection or calculated by the Cockcroft-Gault Formula
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) unless due to Gilbert's disease. For those patients with previous history of Gilbert's disease, a direct bilirubin should be performed and must be <1.5mg/dL.
  * SGOT (AST)/SGPT (ALT) ≤3.0 x the institutional ULN
  * Time from the start of the Q wave to the end of the T wave (QT) corrected for heart rate by Fridericia's cube root formula (QTcF) ≤470 msec

    * For patients with prolonged AT interval due to bundle branch block, a "corrected value" ≤470 msec and confirmation by cardiologist that patient is asymptomatic and that no other cardiac conduction or cardiac abnormality is present would pose any safety issues for the patient.
    * Recommended correction of QT for patients with bundle branch block are as follows: Patient's Q wave R wave and S wave complex (QRS) is 160 msec, and the measured QT is 510 msec. As the normal QRS is ~120 msec, subtract 120 msec from the measured QRS of the patient (160-120 = 40 msec) and then subtract this result from the measured QT (510-40=470 msec).
  * Pulse oximetry reading of ≥90% on room air
* Able to adhere to study visit schedule and other protocol requirements
* Patients must be able to swallow capsules
* Patients must be able to receive xanthine oxidase inhibitor and/or rasburicase for tumor lysis syndrome prophylaxis.
* Patients with a history of hepatitis B (surface antigen or core antibody-positive and polymerase chain reaction (PCR) positive) must take lamivudine or equivalent drug during study therapy and for one year after completion of all therapy. Patients on IVIG who are core antibody-positive but PCR negative are not mandated to take prophylaxis.
* Patients who are HIV (human immunodeficiency virus) positive are eligible under the following circumstances:

  * Undetectable HIV viral load (laboratory value obtained within the last 6 months prior to enrollment)
  * CD4 count ≥200 (laboratory value obtained within the last 6 months prior to enrollment)
  * Actively taking antiretroviral therapy (ART)
  * Current ART therapy cannot have significant interactions with RP-3500 or Olaparib (Refer to Appendix 5). If current medications do interact, patients should receive alternative ART.
* Recovery to baseline or ≤ Grade 1 CTCAE v5.0 from toxicities related to any prior cancer therapy, unless considered clinically not significant by the treating investigator.
* Female patients capable of reproduction or males who have partners capable of reproduction must agree to the use of an effective contraceptive method during the course of the study and for 6 months following the completion of their last treatment.
* Females of childbearing potential must have a negative serum β-Hcg pregnancy test result within 3 days of the first study dose. Female patients who are surgically sterilized or who are >45 years old and have not experienced menses for >2 years may have β-Hcg pregnancy test waived.

Exclusion Criteria:

* Patients who are currently receiving any other investigational drug. Patients who are or have received therapies for the prevention, treatment or management of Corona Virus 19 (COVID-19) under the Food and Drug Administration (FDA) emergency use authorization are allowed to enroll.
* Patients who have received:

  * Radiation or chemotherapy ≤2 weeks prior to registration.
  * Immunotherapy or targeted therapy ≤2 weeks prior to registration.

    ---Patients currently on BCR pathway antagonists (i.e. BTK and PI3K inhibitors, etc) require a 2 day wash out period prior to starting combination therapy with RP-3500 and olaparib as these subjects progress quickly after treatment discontinuation.
  * Strong CYP3A inhibitors or inducers, p-glycoprotein inhibitors, or BCRP inhibitors within five half-lives or 14 days of registration, whichever is shorter (See Appendix 5).
* Prior ATR inhibitor use, but prior PARP inhibitor use for any reason is allowed on study.
* Major surgery 4 weeks prior to C1D1 or who have not fully recovered from major surgery.
* Evidence of active Richter's Transformation
* Disease states requiring steroids (e.g. adrenal insufficiency, autoimmune conditions) are allowed as long as the steroid dose is ≤10mg of prednisone or equivalent dose of another steroid. Steroids premedications to prevent iodine contrast allergy for CT scans are allowed.
* Patients who have undergone autologous stem cell transplant ≤4 weeks or allogeneic stem cell transplant ≤12 weeks prior to cycle 1 day 1 or have active graft-versus-host disease are excluded.
* Patients who have active, clinically significant hepatic impairment (≥ moderate hepatic impairment according to the NCI/Child-Pugh classification)
* Prior history of another malignancy except for the following:

  * Patients with current history of basal or squamous skin carcinoma, cervical carcinoma in situ, localized breast cancer requiring hormonal therapy, or localized prostate cancer (Gleason score <6) are allowed.
  * Previously treated malignancies (with chemotherapy, radiation, and/or surgery) currently deemed to have been in complete remission for at least 24 months.
* Patients with active known central nervous system (CNS) involvement of CLL. Patients with a history of CNS CLL now in remission are eligible for the trial.
* Patients with uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, extensive bilateral interstitial lung disease, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.

  --Patients with a history of pneumonitis or pulmonary disease that could predispose them to development of Interstitial lung disease (ILD) and/or underlying respiratory conditions should be excluded.
* Known prior severe hypersensitivity to RP-3500, olaparib, or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Female patients who are pregnant or actively breast feeding
* Patients with conditions significantly affecting gastrointestinal function including, but not limited to:

  * Significant resection of the stomach or small bowel
  * Symptomatic inflammatory bowel disease
  * Partial or complete bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2025-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boyu Hu, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase Ib: Dose Level -1 | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase II: Dose Expansion Enrichment Cohort | Phase II: Dose Expansion Eligible Subjects Cohort | Phase Ib (Prior to Aug2023 Amendment): Original Dose Level 1
Started | 0 | 0 | 0 | 0 | 0 | 0 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Phase Ib: dose level -1, Phase Ib: dose level 1, Phase Ib: dose level 2, Phase Ib: dose level 3, Phase II: Dose Expansion Enrichment, or Phase II: Dose Expansion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib: Dose Level -1 | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase II: Dose Expansion Enrichment Cohort | Phase II: Dose Expansion Eligible Subjects Cohort | Phase Ib (Prior to Aug2023 Amendment): Original Dose Level 1 | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] |  |  |  |  |  |  | 71.60 (11.60) | 71.60 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  |  |  |  |  | 1 | 1
  Male |  |  |  |  |  |  | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  |  |  |  |  | 0 | 0
  Not Hispanic or Latino |  |  |  |  |  |  | 5 | 5
  Unknown or Not Reported |  |  |  |  |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  |  |  |  |  | 0 | 0
  Asian |  |  |  |  |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  | 0 | 0
  Black or African American |  |  |  |  |  |  | 0 | 0
  White |  |  |  |  |  |  | 5 | 5
  More than one race |  |  |  |  |  |  | 0 | 0
  Unknown or Not Reported |  |  |  |  |  |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  |  |  |  |  |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Camonsertib (RP-3500) in Combination With Olaparib
Description: This outcome will report the number of patients who experienced a Dose-Limiting Toxicity (DLT) in Phase Ib Dose Level 1, Phase Ib Dose Level 2, Phase Ib Dose Level 3, and Phase Ib Dose Level -1 during the DLT window (Cycle 1 Day 1 to Cycle 1 Day 21).
  A keyboard phase I design was employed; the target toxicity was 30% with an equivalence interval between 25-33% of patients. The first 5 patients were treated at DL-1 (camonsertib 40mg daily and olaparib 100mg BID dosing 3 days per week).
Time Frame: up to 28 days after initiation of study drug
Population: No participants were enrolled in the Phase Ib: Dose Level -1, 1, 2, and 3 Cohorts or in the Phase II: Dose Expansion Enrichment or Dose Expansion Cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Dose Level -1 | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase II: Dose Expansion Enrichment Cohort | Phase II: Dose Expansion Eligible Subjects Cohort | Phase Ib (Prior to Aug2023 Amendment): Original Dose Level 1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5
Participants
  Experienced a DLT |  |  |  |  |  |  | 1
  Did not Experience a DLT |  |  |  |  |  |  | 4
Statistical Analysis 1: Comparison: Phase Ib: Dose Level -1; Test type: Other; The primary analysis was of safety and included all patients who received at least one dose of the investigational regimen. The rate of adverse events was estimated after the first 5 patients were treated at Original DL1 (camonsertib 40mg daily and olaparib 100mg BID dosing 2 days per week, at 28 day cycles) After the first 5 patients were treated, it was determined that this dosing strategy may not be appropriate for R/R CLL patients and reduced dosing frequency may be necessary to increase the safety of the combination therapy. The protocol and DLs were amended, and sought to enroll an additional 18 patients. Before the enrollment of 18 additional participants and MTD determination, the study was terminated due to sponsor de-activation of all programs associated with camonsertib

2. Primary Outcome: Overall Response
Description: This outcome will assess the overall responseof combination RP-3500 and olaparib. Overall response is defined by the count of subjects achieving any confirmed partial (PR) and complete response (CR) as assessed by 2018 International Working Group on Chronic Lymphocytic Leukemia (iwCLL) response criteria.
  Subjects without a baseline/screening tumor assessment or at least one on-treatment assessment will be considered non-responders.
Time Frame: up to 85 Days after initiation of study drug
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Dose Level -1 | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase II: Dose Expansion Enrichment Cohort | Phase II: Dose Expansion Eligible Subjects Cohort | Phase Ib (Prior to Aug2023 Amendment): Original Dose Level 1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5
Participants |  |  |  |  |  |  | 0

3. Secondary Outcome: Adverse Events (AE) by Grade
Description: This outcome measure will assess the safety and tolerability of RP-3500 and olaparib.
  The severity of AEs was assessed using CTCAE v5.0 criteria, a 1-5 scale with higher numbers indicating greater severity. Grade 1 indicates "mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated" and Grade 5 indicates "death related to AE".
  The severity of adverse hematologic adverse events was assessed using the 2018 IWCLL grading scale. Grade 0 indicates "≤10% decrease in platelets (PLT) or hemoglobin (Hb) from baseline and ≥2 absolute neutrophil count (ANC)" and Grade 4 indicates "≥75% decrease in PLT or Hb from baseline and <0.5 ANC"
  This outcome measure will report the count of participants who experienced each AE grade. Subjects were monitored for adverse events from the start of treatment until 28 days after the last dose of the study drug.
Time Frame: up to 28 days after the last dose of study treatment (up to 113 days after initiation of study drug)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Dose Level -1 | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase II: Dose Expansion Enrichment Cohort | Phase II: Dose Expansion Eligible Subjects Cohort | Phase Ib (Prior to Aug2023 Amendment): Original Dose Level 1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5
Participants
  CTCAE Grade 1 | 0 |  |  |  |  |  | 4
  CTCAE Grade 2 | 0 |  |  |  |  |  | 3
  CTCAE Grade 3 | 0 |  |  |  |  |  | 3
  CTCAE Grade 4 | 0 |  |  |  |  |  | 1
  CTCAE Grade 5 |  |  |  |  |  |  | 0
  iwCLL Hematologic Grade 0 |  |  |  |  |  |  | 0
  iwCLL Hematologic Grade 1 |  |  |  |  |  |  | 0
  iwCLL Hematologic Grade 2 |  |  |  |  |  |  | 0
  iwCLL Hematologic Grade 3 |  |  |  |  |  |  | 4
  iwCLL Hematologic Grade 4 |  |  |  |  |  |  | 3

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) as defined as the time from study drug initiation to the time documented disease progression (as assessed by 2018 iwCLL criteria) or death from any cause. Patients were followed for PFS until progression of disease was noted or death, whichever occurred first.
  This outcome will report the median PFS with 95% confidence intervals.
Time Frame: up to 15 months from initiation of study treatment
Population: No participants were enrolled in the Phase Ib: Dose Level 1, 2, and 3 Cohorts or in the Phase II: Dose Expansion Enrichment or Dose Expansion Cohorts.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib: Dose Level -1 | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase II: Dose Expansion Enrichment Cohort | Phase II: Dose Expansion Eligible Subjects Cohort | Phase Ib (Prior to Aug2023 Amendment): Original Dose Level 1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5
months |  |  |  |  |  |  | 2.66 [0 to 9.33]

5. Secondary Outcome: Overall Survival (OS)
Description: This outcome will assess OS as defined as the time between treatment initiation and death of any cause.
  Subjects were followed for OS from the initiation of therapy until death from any cause or until the study was terminated. Subjects lost to follow-up or refused follow-up were censored at the time of the last known follow-up.
  This outcome will report the median OS with 95% confidence intervals.
Time Frame: up to 21 months after study registration
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib: Dose Level -1 | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase II: Dose Expansion Enrichment Cohort | Phase II: Dose Expansion Eligible Subjects Cohort | Phase Ib (Prior to Aug2023 Amendment): Original Dose Level 1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5
months |  |  |  |  |  |  | 14.70 [0 to 56.06]

6. Secondary Outcome: Duration of Response (DoR) as Defined as the Interval of Time From the Date of Initial Documented Response (PR or Better as Per 2018 iwCLL Criteria for Response) to the Time of Progression.
Description: DoR is defined as the interval of time from the date of the initial documented response (PR or better as per 2018 iwCLL criteria for response) to the time of progression.
  Patients would be followed for DoR from the date of the initial documented response until progression of disease was noted or death, whichever occurred first.
  This outcome would have reported the median DoR with 95% confidence intervals.
Time Frame: up to 21 months after initiation of study treatment.
Population: No participants had an initial documented response.
Arm/Group | Phase Ib: Dose Level -1 | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase II: Dose Expansion Enrichment Cohort | Phase II: Dose Expansion Eligible Subjects Cohort | Phase Ib (Prior to Aug2023 Amendment): Original Dose Level 1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events from the start of treatment until 28 days after the last dose of the study drug (up to 113 days after initiation of study drug). Subjects were monitored for survival for up to 21 months after study registration.
Description: No participants were enrolled in the Phase Ib: Dose Level 1, 2, and 3 Cohorts or in the Phase II: Dose Expansion Enrichment or Dose Expansion Cohorts.
Groups:
- Phase Ib: Dose Level -1: To assess the MTD of RP-3500 in combination with olaparib. Patients will receive 40mg of RP-3500 daily and 100mg Olaparib BID.
  RP-3500: RP-3500 is a highly potent and selective Ataxia telangiectasia and Rad3 related inhibitor (ATRi) and has demonstrated significant preclinical activity.
  Olaparib: Olaparib is an oral poly (adenosine diphosphate-ribose) polymerase inhibitor (PARPi) that inhibits PARP's function by competitively binding to the Nicotinamide adenine dinucleotide (NAD+) binding site, which PARP requires as a cofactor to operate.
- Phase Ib: Dose Level 1: To assess the MTD of RP-3500 in combination with olaparib. Patients will receive 50mg of RP-3500 daily and 100mg Olaparib BID.
  RP-3500: RP-3500 is a highly potent and selective Ataxia telangiectasia and Rad3 related inhibitor (ATRi) and has demonstrated significant preclinical activity.
  Olaparib: Olaparib is an oral poly (adenosine diphosphate-ribose) polymerase inhibitor (PARPi) that inhibits PARP's function by competitively binding to the Nicotinamide adenine dinucleotide (NAD+) binding site, which PARP requires as a cofactor to operate.
- Phase Ib: Dose Level 2: To assess the MTD of RP-3500 in combination with olaparib. Patients will receive 80mg of RP-3500 daily and 100mg Olaparib BID.
  RP-3500: RP-3500 is a highly potent and selective Ataxia telangiectasia and Rad3 related inhibitor (ATRi) and has demonstrated significant preclinical activity.
  Olaparib: Olaparib is an oral poly (adenosine diphosphate-ribose) polymerase inhibitor (PARPi) that inhibits PARP's function by competitively binding to the Nicotinamide adenine dinucleotide (NAD+) binding site, which PARP requires as a cofactor to operate.
- Phase Ib: Dose Level 3: To assess the MTD of RP-3500 in combination with olaparib. Patients will receive 80mg of RP-3500 daily and 150mg Olaparib BID.
  RP-3500: RP-3500 is a highly potent and selective Ataxia telangiectasia and Rad3 related inhibitor (ATRi) and has demonstrated significant preclinical activity.
  Olaparib: Olaparib is an oral poly (adenosine diphosphate-ribose) polymerase inhibitor (PARPi) that inhibits PARP's function by competitively binding to the Nicotinamide adenine dinucleotide (NAD+) binding site, which PARP requires as a cofactor to operate.
Arm/Group | Phase Ib: Dose Level -1 | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase II: Dose Expansion Enrichment Cohort | Phase II: Dose Expansion Eligible Subjects Cohort | Phase Ib (Prior to Aug2023 Amendment): Original Dose Level 1
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 2/5
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 2/5
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib: Dose Level -1 (N=0) | Phase Ib: Dose Level 1 (N=0) | Phase Ib: Dose Level 2 (N=0) | Phase Ib: Dose Level 3 (N=0) | Phase II: Dose Expansion Enrichment Cohort (N=0) | Phase II: Dose Expansion Eligible Subjects Cohort (N=0) | Phase Ib (Prior to Aug2023 Amendment): Original Dose Level 1 (N=5)
Anemia (Blood and lymphatic system disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Urinary tract infection (Infections and infestations) | NA | NA | NA | NA | NA | NA | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib: Dose Level -1 (N=0) | Phase Ib: Dose Level 1 (N=0) | Phase Ib: Dose Level 2 (N=0) | Phase Ib: Dose Level 3 (N=0) | Phase II: Dose Expansion Enrichment Cohort (N=0) | Phase II: Dose Expansion Eligible Subjects Cohort (N=0) | Phase Ib (Prior to Aug2023 Amendment): Original Dose Level 1 (N=5)
Anemia (Blood and lymphatic system disorders) | NA | NA | NA | NA | NA | NA | 1 (3)
Anorexia (Metabolism and nutrition disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Bruising (Injury, poisoning and procedural complications) | NA | NA | NA | NA | NA | NA | 2 (2)
Constipation (Gastrointestinal disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Creatinine increased (Investigations) | NA | NA | NA | NA | NA | NA | 1 (3)
Diarrhea (Gastrointestinal disorders) | NA | NA | NA | NA | NA | NA | 2 (2)
Dizziness (Nervous system disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Dyspepsia (Gastrointestinal disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Edema limbs (General disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Fall (Injury, poisoning and procedural complications) | NA | NA | NA | NA | NA | NA | 1 (1)
Fatigue (General disorders) | NA | NA | NA | NA | NA | NA | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Headache (Nervous system disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | NA | NA | NA | NA | NA | NA | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | NA | NA | NA | NA | NA | NA | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | NA | NA | NA | NA | NA | NA | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | NA | NA | NA | NA | NA | NA | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Lung infection (Infections and infestations) | NA | NA | NA | NA | NA | NA | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | NA | NA | NA | NA | NA | NA | 1 (2)
Nausea (Gastrointestinal disorders) | NA | NA | NA | NA | NA | NA | 3 (3)
Neutrophil count decreased (Investigations) | NA | NA | NA | NA | NA | NA | 2 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Platelet count decreased (Investigations) | NA | NA | NA | NA | NA | NA | 3 (9)
Sepsis (Infections and infestations) | NA | NA | NA | NA | NA | NA | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | NA | NA | NA | NA | NA | NA | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Tinnitus (Ear and labyrinth disorders) | NA | NA | NA | NA | NA | NA | 1 (1)
Urinary tract infection (Infections and infestations) | NA | NA | NA | NA | NA | NA | 1 (1)
Weight loss (Investigations) | NA | NA | NA | NA | NA | NA | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT05405309/Prot_SAP_000.pdf